CLINICAL TRIAL: NCT03707769
Title: First-in-human Open Label Feasibility Study to Assess the Safety of TIPS Microspheres in Perianal Fistulas
Brief Title: TIPS Microspheres for Perianal Fistula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14/0845
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Perianal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fistula treatment (Experimental): Treatment of fistula with TIPS microspheres
  Interventions: Device: TIPS microspheres

INTERVENTIONS:
Device: TIPS microspheres — TIPS microspheres manufactured from GMP grade poly(lactide-co-glycolide) (PLGA) prepared as a paste with GranuGel.

SUMMARY:
Phase of Investigation: First-in-human feasibility study

Objectives: Primary objective: Demonstration that TIPS microspheres do not compromise the clinical condition or safety of the patient.

Secondary objective: To demonstrate that TIPS microspheres facilitate natural healing in the context of perianal fistula.

Type of Investigation: First-in-human single site, open label, feasibility study to assess the safety of TIPS microspheres in perianal fistulas and indicative functionality.

Investigation design and methods: First-in-human single delivery of a bioabsorbable device to treat perianal fistula. A standard of care internal flap procedure performed to close the internal fistula opening and up to 300 mg of TIPS microspheres will be inserted into each perianal fistula. Participants will be assessed for healing, inflammation, abscess, sepsis, pain and continence by clinical assessments, blood tests, MRI and questionnaires.

DETAILED DESCRIPTION:
TIPS microspheres are manufactured from GMP grade poly(lactide-co-glycolide) (PLGA) under Good Laboratory Practice (GLP) conditions.

Microspheres will be delivered into the fistula tract using the following procedure:

i) Tract identification with special emphasis on locating the internal and external openings using a fistula probe.

ii) Curettage to remove epithelium lining the tract and cleaning by irrigation with hydrogen peroxide and saline.

iii) Closure of the internal opening by means of a rectoanal advancement flap. iv) Following device kit instructions, prepare a paste of TIPS microspheres with GranuGel.

v) Introduction of TIPS microsphere paste by back-filling. vi) Retention of the microsphere paste using Comfeel adhesive hydrocolloid dressing designed to remain in place for 1 - 14 days.

Each subject will receive a single administration of up to 300 mg of TIPS microspheres implanted into the fistula tract.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* Cryptoglandular perianal fistula
* High and low simple trans-sphincteric fistula

Exclusion Criteria:

* Secondary fistula, including Crohn's disease, carcinoma, radiotherapy, tuberculosis
* Evidence of branching fistula anatomy or cavity on MRI
* Inter-sphincteric fistula
* Low trans-phincterictrans-sphincteric fistula amenable to simple fistulotomy
* Immunosuppressed patients
* Participants less than 18 years of age
* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Within 9 months of device implantation
  Safety as defined by morbidity, measured by occurrence of adverse events / reactions, in particular: perianal sepsis, perianal abscess, or reoperation due to sepsis

SECONDARY OUTCOMES:
Clinical evidence of fistula healing | 9 months after device implantation
  Efficacy through facilitation of natural healing as determined by: clinical evidence of fistula healing; MRI evidence of fistula healing; improvement of quality of life assessment Improvement of pain score assessment

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospitals, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No